CLINICAL TRIAL: NCT06955962
Title: Examining the Effect of Mandala Art Therapy on Symptoms and Quality of Life in Multiple Sclerosis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Müge TEZEL, Research assistant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MTEZEL
Record Dates: First submitted 2025-04-11; First posted 2025-05-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mandala art therapy; quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The mandala art therapy for individuals in the intervention group is planned to be conducted in their home environments under suitable conditions. The therapy sessions will be accompanied by music of the participants' choosing and are scheduled to take place over a six-week period, at least three to four times per week, for a minimum of 30 minutes per session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In the study, no intervention will be applied to individuals in the control group during their visits to the neurology outpatient clinic; they will continue with their routine follow-up, examinations, and treatment as usual. Pre-tests will be administered to participants in the control group who agree to take part in the study, have been informed about its purpose, scope, duration, and methodology, and have provided both written and verbal consent. These pre-tests will include the "Descriptive Information Form," the "Multiple Sclerosis Symptom Scale (MS-RS)," and the "Multiple Sclerosis Quality of Life Scale (MSQL-54)."
  At the end of six weeks, participants will be contacted via telephone to schedule an appointment for the administration of post-tests. The post-tests to be applied to the control group will again include the "Descriptive Information Form," the "Multiple Sclerosis Symptom Scale (MS-RS)," and the "Multiple Sclerosis Quality of Life Scale (MSQL-54)."
- Intervention Group (Experimental): The mandala art therapy for individuals in the intervention group is planned to be conducted in their home environments under suitable conditions. The therapy sessions will be accompanied by music of the participants' choosing and are scheduled to take place over a six-week period, at least three to four times per week, for a minimum of 30 minutes per session.
  Interventions: Other: Mandala Art Therapy

INTERVENTIONS:
Other: Mandala Art Therapy — Arm Description: The mandala art therapy for individuals in the intervention group is planned to be conducted in their home environments under suitable conditions. The therapy sessions will be accompanied by music of the participants' choosing and are scheduled to take place over a six-week period, at least three to four times per week, for a minimum of 30 minutes per session. Before the first mandala art therapy session, participants in the intervention group will receive a brief orientation by the researcher on the appropriate environment for the practice and an introduction to mandala art therapy. This orientation will include information on the definition and characteristics of mandala art therapy, the application setting and duration, and general guidelines to be followed during the sessions. At the end of the six-week mandala art therapy program, Post-tests ill be administered face-to-face, and the archived mandala folders will be collected
  Arms: Intervention Group

SUMMARY:
This study is a randomized controlled, pre-test-post-test experimental research aimed at examining the effects of mandala art therapy on symptom severity and quality of life in individuals diagnosed with Multiple Sclerosis (MS). The main goal is to determine whether mandala art therapy helps reduce the frequency and severity of MS symptoms while improving participants' overall quality of life.

It is expected that mandala art therapy will support MS patients in managing current and potential symptoms, coping more effectively with the disease, and improving adherence to treatment. As a result, a reduction in healthcare utilization, related costs, MS-related complications, and mortality is anticipated.

The study will be conducted between May and August 2025 at the Neurology Outpatient Clinic of Karadeniz Technical University Practice and Research Center, involving 70 patients-35 in the intervention group receiving mandala art therapy and 35 in the control group receiving standard care.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled, pre-test-post-test experimental research to examine the effects of mandala art therapy on symptom severity and quality of life in individuals diagnosed with Multiple Sclerosis (MS). The primary objective of the study is to evaluate whether the implementation of mandala art therapy contributes to a reduction in the frequency and severity of MS-related symptoms, while simultaneously enhancing the overall quality of life of the participants.

In this context, it is anticipated that mandala art therapy may support individuals with MS in managing existing and potential symptoms, coping more effectively with the disease, and achieving better adherence to treatment and disease management. Consequently, it is expected that the frequency of healthcare utilization and overall healthcare-related costs will decrease. Most importantly, a reduction in MS-related complications and mortality is also anticipated.

The planned study will be conducted between May 2025 and August 2025 at the Neurology Outpatient Clinic of the Karadeniz Technical University Practice and Research Center, involving a total of 70 patients-35 in the intervention group and 35 in the control group-who meet the inclusion criteria. While patients in the intervention group will receive mandala art therapy, those in the control group will continue their routine follow-up and treatment without any additional intervention.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the city center of Trabzon
* Diagnosed with Multiple Sclerosis at least six months prior
* Have not experienced an MS relapse within the past three months
* Receiving outpatient treatment for MS
* Literate
* Have no prior experience with mandala practice
* Not currently participating in any form of art therapy
* Have no communication or perception impairments

Exclusion Criteria:

* Those who have experienced an MS relapse within the past three months
* Those receiving inpatient treatment for MS
* Individuals aged 18 years or younger
* Those with a physical disability that prevents them from participating in the mandala activity
* Individuals currently engaged in any form of active art therapy
* Those with communication or perception impairments
* Individuals with a diagnosed psychiatric disorder
* Those who cannot be reached via phone and/or text message
* Individuals with allergies to materials used in the mandala therapy sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patient with MS | 6 week
  The quality of life of patient with MS will be defined by using Multiple Sclerosis Quality of Life Scale (MSQL-54).
  The scale scores range from 0 to 100, and as the score increases, the quality of life of individuals increases.

SECONDARY OUTCOMES:
Symptom evaluation of patient with MS | 6 week
  Symptom evaluation of patient with MS will be defined by using Multiple Sclerosis Symptom Scale (MS-RS) The minimum score that can be obtained from the scale is 0, the maximum score is 130, with higher scores indicating increased symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin NURAL, Prof, Study Director — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This thesis study is currently ongoing and has not yet been completed.